CLINICAL TRIAL: NCT06497309
Title: Advanced Technology-based Rehabilitation Programmes to Support Gait Re-learning After Stroke
Brief Title: Advanced Technology-based Rehabilitation Post-stroke Gait Re-learning
Status: Enrolling by invitation | Type: Observational
Sponsor: National Institute for Medical Rehabilitation, Hungary (Other Government)
Collaborators: Semmelweis University (Other)
Responsible Party: Sponsor
Other Study IDs: OMINT-58-1/2023
Record Dates: First submitted 2024-04-03; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-05

CONDITIONS: Stroke; Gait Disorders, Neurologic
Keywords: Rehabilitation; Physical Therapy; High-tech devices; Stroke; Gait re-learning
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treadmill group: In both groups, using advanced technology-based tools (both treatments are part of the daily routine of the Institute's treatments and are used according to the instructions in the user manual), for the treadmill therapy, we use the C-Mill interactive high-tech device.
  Interventions: Device: Treadmill training; Device: DIERS; Other: Traditional physiotherapy assessments
- Overground group: In both groups, we use an advanced technology-based device (both treatments are part of the daily routine of the Institute's treatments and are used according to the instructions in the user manual), and the Andago high-tech device for non-runner therapy.
  Interventions: Device: Overground training; Device: DIERS; Other: Traditional physiotherapy assessments

INTERVENTIONS:
Device: Treadmill training — Therapy with treadmill-based advanced technology device.
  Groups: Treadmill group
Device: Overground training — Therapy using an advanced technological device enables exercise on the ground.
  Groups: Overground group
Device: DIERS — The examination starts and ends with the DIERS motion analysis system, a light-optical scanning method based on VRS (Video Raster Stereography) and a sensor-equipped treadmill that allows the measurement of several parameters of gait and balancing ability.
Other: Traditional physiotherapy assessments — Traditional physiotherapy assessment methods (Timed Up and Go, Berg Balance Test, 6-minute gait test, 10-metre gait test, Functional Independence Measure, Barthel) are used to assess gait pattern and self-sufficiency.

SUMMARY:
High-tech therapy, an innovative field of neurorehabilitation, has expanded rapidly in recent years. Advances in technology have enabled the use of devices that can assist with movement development from simple movements to more complex tasks.

This research investigates the effectiveness of rehabilitation programmes that complement robot-assisted therapy to help people relearn to walk in post-stroke rehabilitation. This would be measured in two variations, with the patient (in addition to a complex rehabilitation programme of conventional physiotherapy, occupational therapy, hydrotherapy, etc.) receiving either treadmill or no treadmill treatment. In both cases, the therapies will be carried out with advanced technology-based equipment (both treatments are part of the daily routine of the Institute's treatments, and the equipment will be used according to the instructions in the user manual), the C-Mill interactive robot-assisted device will be used for treadmill therapy, and the Andago robot-assisted device for non- treadmill therapy. There is no sharp distinction between the two systems. The inclusion and exclusion criteria are set so patients' conditions meet the indications for both devices, and patients eligible for treatment with one device are included in the other.

In our study, 80 patients will be selected.

DETAILED DESCRIPTION:
The main objective of this research is to investigate the effectiveness of rehabilitation programmes in post-stroke rehabilitation using advanced technology-based therapy to assist in relearning walking. This will be measured in two variations: the patient will be randomly assigned (in addition to a complex rehabilitation programme of traditional physiotherapy, occupational therapy, hydrotherapy, etc.) to receive either treadmill treatment or no treadmill treatment. In both cases, the therapies are carried out using advanced technological equipment.

The investigators will enrol 80 people in our study. The comparison will be between 40 and 40 people, the main groups differing in terms of the type of advanced technology device used in the rehabilitation programme and whether they received treadmill or non-treadmill treatment. In total, they will participate in 20 sessions of therapy.

Furthermore, the investigators observe whether a greater change in condition can be measured in the early post-stroke period (0-3 months) or the late period (3 months-1 year) in specific parameters of the patient's gait. The time since the stroke provides an opportunity for subgroup analysis, but the number of cases limits this. This is significant because it is still an open question in the international literature regarding advanced technology-based therapy.

In all cases, the examination starts and ends with the DIERS motion analysis system, a light-optical scanning method based on VRS (Video Raster Stereography) and a sensor-equipped treadmill that allows the measurement of several parameters of gait and balancing ability. In addition, traditional physiotherapy assessment methods (Timed Up and Go, Berg Balance Test, 6-minute gait test, 10-metre gait test, Functional Independence Measure, Barthel) are used to assess gait pattern and self-sufficiency.

ELIGIBILITY:
Inclusion Criteria:

* Hemiparetic patient who has had a stroke;
* ischaemic or haemorrhagic stroke confirmed by CT or MRI;
* female or male between 40 and 75 years of age;
* subgroup 1: less than 3 months since stroke,
* subgroup 2: more than 3 months but less than 1 year since stroke;
* physical fitness adequate for the exertion of the treatment;
* right or left lower limb involvement;
* score 3 on the Functional Ambulation Categories (FAC) scale, i.e. Indicates a patient who can ambulate on a level surface without manual contact of another person but requires standby guarding of one person either for safety or verbal cueing;
* or score 4 on the Functional Ambulation Categories (FAC) scale, i.e. Indicates a patient who can ambulate independently on a level surface but requires supervision to negotiate (e.g. stairs, inclines, non-flat surfaces);
* be able to participate in therapy and cooperate based on cognitive function;
* signed informed consent.

Exclusion Criteria:

* More than 1 year has passed since the stroke;
* scores less than or equal to 3 on the Functional Ambulation Categories (FAC) scale;
* patients who were unable to walk independently before the stroke;
* patients treated with botulinum toxin in the lower limb in the last 3 months;
* use of other lower limb advanced technology treatments during the study;
* a person with limited capacity;
* not physically able to bear weight;
* severe aphasia (impairment of understanding or expression that severely impedes communication);
* other condition that precludes the use of C-Mill or Andago:

  * severe emotional disturbance;
  * mentally incapacitated patient;
  * severe contracture or spasticity preventing the patient from being placed in the machine;
  * pregnancy;
  * skin disease in the area of contact with the straps;
  * fever;
  * unhealed fracture fracture;
  * inability to use the device due to weight and height limitations of the device;
  * epilepsy if you have had a seizure within a year;
  * severe visual impairment.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the National Institute for Medical Rehabilitation, Budapest, Hungary
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Balancing skills | Through study completion, an average of 2 years.
  Berg Balance Test (values between 0-56, higher score means better outcome).
Balancing skills | Through study completion, an average of 2 years.
  Timed Up and Go Test (how many seconds it takes the patient to complete the task).
Balancing skills | Through study completion, an average of 2 years.
  Weight distribution (%) using the DIERS medical device.
Balancing skills | Through study completion, an average of 2 years.
  COP movement (mm) using the DIERS medical device.
Balancing skills | Through study completion, an average of 2 years.
  Sway area (mm2) using the DIERS medical device.
Balancing skills | Through study completion, an average of 2 years.
  Romberg opened eyes, closed eyes (mm) using the DIERS medical device.
Balancing skills | Through study completion, an average of 2 years.
  Strength of the lower limbs (hip extension, flexion, adduction and abduction) and the trunk (flexion, extension, rotation, lateroflexion) (N) using the DIERS medical device.
Gait parameters | Through study completion, an average of 2 years.
  6-minute gait test (m).
Gait parameters | Through study completion, an average of 2 years.
  10-meter gait test (min).
Gait parameters | Through study completion, an average of 2 years.
  step length (mm), using the DIERS medical device.
Gait parameters | Through study completion, an average of 2 years.
  Step width (mm), using the DIERS medical device.
Gait parameters | Through study completion, an average of 2 years.
  Heel strike (N), using the DIERS medical device.
Gait parameters | Through study completion, an average of 2 years.
  COP movement (mm), using the DIERS medical device.
Functional independence | Through study completion, an average of 2 years.
  Based on FIM (maximum 126 points, higher score means better outcome).
Functional independence | Through study completion, an average of 2 years.
  Based on Barthel (values between 0-99, higher score means better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Gábor Fazekas, MD, PhD, Principal Investigator — National Institute for Medical Rehabilitation, Hungary
Locations (1):
- National Institute for Medical Rehabilitation, Budapest, Pest County, Hungary